CLINICAL TRIAL: NCT02936310
Title: Effect of Mindful Living With Stress (MLWS) Intervention for Nurses Caring for HIV/AIDS Patients in China
Brief Title: Mindful Living With Stress for Nurses Caring for HIV/AIDS Patients in China
Acronym: MLWS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Chen Pan, Dr., Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16-001305
Record Dates: First submitted 2016-10-13; First posted 2016-10-18 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Stress
Keywords: stress; mindfulness; Mindful Living With Stress Intervention; nurse; HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mindfulness intervention (Experimental): The proposed Mindful Living With Stress Intervention will be conducted weekly, 2 hours per session, 4-6 sessions, group based program in mindfulness.The proposed topics include: 1) mindfulness: dealing with stress in a new way, 2) mindful awareness of stress: listening to our body, 3) mindful working with thoughts, 4) mindful working with emotions, 5) mindful interactions, and 6) dealing with obstacles of mindful practices and wrap-up. Mindfulness practices embedded in the program will include mindfulness breathing meditation, sitting meditation, standing meditation, walking meditation, movement meditation (Taichi or Yoga), body scan meditation and daily life meditation.
  Data will be collected at pre-intervention (one week before the first session) and post-intervention (one week after the last session) to assess stress, burnout, mindfulness, anxiety,depression,the feedback on the MLWS intervention and the feedback on the influence of MLWS intervention.
  Interventions: Behavioral: Mindful Living With Stress

INTERVENTIONS:
Behavioral: Mindful Living With Stress — The proposed Mindful Living With Stress Intervention will be conducted weekly, 2 hours per session, 4-6 sessions, group based program in mindfulness.

SUMMARY:
The primary objective of this proposed one-year (January 01, 2017 to December 31,2017) project is to assess whether a mindfulness based intervention('Mindful Living With Stress') will be effective at helping nurses caring for HIV/AIDS patients in China to reduce stress. Based on the efficacy of previous studies in stress reduction, it is hypothesized that 'Mindful Living With Stress' will be an effective, feasible and affordable stress reduction program in China.

DETAILED DESCRIPTION:
Background: Considering the great stress in the nurses caring for HIV/AIDS patients, the situation of more serious nursing shortage in China, and the acceptability, feasibility and efficacy of mindfulness-based interventions for reducing stress in health care professionals, here investigators propose a study of "Effect of Mindful Living With Stress (MLWS) Intervention for nurses caring for HIV/AIDS patients in China".

Objectives: The primary objective of this proposed project is to assess whether a program of mindfulness-based stress reduction interventions developed based on Mindfulness Based Stress Reduction (MBSR), Mindful Awareness Practices（MAPs）and chinese culture will be effective at helping nurses caring for HIV/AIDS patients in China to reduce stress and burnout. Based on the efficacy of previous studies in reducing stress, investigators hypothesize that 'Mindful Living With Stress' will be an effective, feasible and affordable stress reduction program for nurses caring for HIV/AIDS patients in China.

Methods: Nurses working in the AIDS department of the First Hospital of Changsha, China will be recruited for the study. The two steps to be implemented include: 1) conducting focus groups with nurses for the purpose of finalizing the design of the MLWS Intervention: A convenience sample of 10 nurses will be recruited and the final sample is expected to include 6-8 participants who will attend two consecutive focus group sessions. The first focus group session will explore the experiences of nurses caring for HIV/AIDS patients and the second focus group session will discuss the design of the MLWS Intervention. The qualitative data will be analyzed after the focus group discussions and the findings will provide important information for development of the final manual for guiding the intervention, and 2) evaluating the effects of the MLWS Intervention in a group of nurses: A convenience sample of 23 nurses will be recruited and the final sample is expected to include 16-18 nurses. The quantitative data from 5 measures assessing stress, burnout, mindfulness, anxiety and depression will be collected and analyzed at pre- and post- intervention. The qualitative data from an in-depth interview will be collected and analyzed at post-intervention.

Implications: The results will provide valuable insights into the effect of MLWS Intervention on stress of nurses caring for HIV/AIDS patients in China. If the MLWS Intervention can be used effectively, it can also be popularized to many other health care professionals caring for HIV/AIDS in China in future.

ELIGIBILITY:
The first step of the study:focus group

Inclusion Criteria:

1. having a license to practice as a nurse in the People's Republic of China.
2. being employed as a nurse in the AIDS department of the First Hospital of Changsha for at least 1 year.
3. Chinese speaking.
4. being at least 18 years old.

Exclusion Criteria:

1. being other types of health care providers such as doctors, pharmacists, social workers.
2. being a nursing supervisor or manager.

The second step of the study: mindfulness intervention

Inclusion Criteria:

1. having a license to practice as a nurse in the People's Republic of China.
2. being employed as a nurse in the AIDS department of the First Hospital of Changsha for at least 1 year.
3. Chinese speaking.
4. being at least 18 years old.

Exclusion Criteria:

1. being other types of health care providers such as doctors, pharmacists, social workers.
2. being a nursing supervisor or manager.
3. having attended in the focus group of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
stress assessed with a self-administrated questionnaire （Chinese Version of Perceived Stress Scale） | nine month
  At the pre- and post-intervention assessment, participants will complete self-administrated questionnaire on stress.
stress assessed with an in-depth interview | nine month
  At the post-intervention assessment,participants will be invited to attend an in-depth interview to give the feedback on the influence of MLWS intervention on living with stress.

SECONDARY OUTCOMES:
burnout assessed with a self-administrated questionnaire (Chinese Version of Maslach Burnout Inventory) | nine month
mindfulness assessed with a self-administrated questionnaire (Chinese Version of Five Facets Mindfulness Questionnaire) | nine month
anxiety assessed with a self-administrated questionnaire （State-Trait Anxiety Inventory） | nine month
depression assessed with a self-administrated questionnaire （Beck Depression Inventory） | nine month

CONTACTS AND LOCATIONS:
Overall Officials: Chen Pan, M.D., Ph.D., Principal Investigator — Central South University
Locations (1):
- The First Hospital of Changsha, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
data will be made available within 6 months of study completion